CLINICAL TRIAL: NCT05642273
Title: The Effects of extraCorporeal bLood Purification (oXiris ®) in patiEnts With cArdiogeNic Shock Requiring VA-ECMO: A Prospective, Open-label, Randomized Controlled Pilot Study
Brief Title: The Effects of oXiris in Cardiogenic Shock Requiring VA-ECMO
Acronym: CLEAN ECMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Hoon Yang, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLEAN ECMO
Record Dates: First submitted 2022-11-28; First posted 2022-12-08 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Cardiogenic Shock
Keywords: cardiogenic shock; venoarterial extracorporeal membrane oxygenation; endotoxin; cytokine; oXiris
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Oxiris for 24 h
  Interventions: Device: oXiris membrane; Diagnostic Test: Blood tests
- Control (Active Comparator): Usual care
  Interventions: Diagnostic Test: Blood tests

INTERVENTIONS:
Device: oXiris membrane — oXiris membrane for 24h
  Arms: Intervention
Diagnostic Test: Blood tests — Blood tests just after randomization (0 h) and at 24 h, 48 h and 7 days

SUMMARY:
Cardiogenic shock (CS) defines a state of systemic hypo-perfusion leading to end-organ dysfunction related to cardiac pump failure and with mortality rates in the range of 27-50% according to recent reviews. Patients with CS often received mechanical circulatory support, and venoarterial extracorporeal membrane oxygenator (V-A ECMO) is an effective tool to support refractory CS while ensuring continuous organ perfusion. Patients with CS present clinical signs of systemic inflammation and elevated plasma levels of prototypical inflammatory and vasoactive mediators, including C-reactive protein (CRP), Interleukin-6 (IL-6) and tumor necrosis factor alpha (TNFα). As data is scarce in this field, we decided to perform a prospective randomized controlled pilot study to investigate the efficacy of extracorporeal cytokine and lipopolysaccharide adsorption using Oxiris on humoral inflammation parameters, hemodynamics, and clinical outcomes in patients with CS requiring VA ECMO.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with more than 18 years old
2. CS is defined as the presence of the following:

   2-1) Systolic blood pressure is less than 90 mmHg for more than 30 minutes despite the fluid therapy, or the use of pressure boosting agents to maintain the systolic blood pressure more than 90 mmHg.

   2-2) Peripheral hypoperfusion (cold skin, urine less than 30 cc per hour, impaired consciousness, lactate ≥2.0 mmol/l) or a person with pulmonary edema.

   2-3) Causes of CS include ischemic (acute myocardial infarction or ischemic cardiomyopathy, shock during percutaneous coronary intervention), myocardial (end-stage heart failure, myocarditis), post-cardiotomy shock, cardiac tamponade, or pulmonary thromboembolism.
3. Patients receiving VA ECMO owing related to the causes listed in 2-1, 2-2, 2-3.
4. Written informed consent from patient or legal surrogates

Exclusion Criteria:

1. Other causes except for CS: septic shock, cardiac arrest by serious ventricular arrhythmia mot related to the myocardial ischemia or heart failure.
2. Shock with unwitnessed cardiac arrest outside the hospital
3. Severe non-cardiac morbidity with expected survival less than 6 months (malignancy, respiratory failure)
4. Suspicious of brain death
5. Those who refused active treatment
6. Body weight under 30 kg
7. Heparin allergy
8. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Endotoxin level at 48 h | 48 hours after enrollment
  Plasma endotoxin level

SECONDARY OUTCOMES:
Vasoactive-Inotrope score | baseline, 24 hours, 48 hours, 72 hours, 96 hours, Day 7
  VIS = dopamine (µg/kg/min) + dobutamine (µg/kg/min) + 100 × epinephrine (µg/kg/min) + 100 × norepinephrine (µg/kg/min) + 10 × milrinone (µg/kg/min) + 10,000 × vasopressin (units/kg/min) + 50 × levosimendan (µg/kg/min)
Sequential Organ Failure Assessment score | baseline, 24 hours, 48 hours, 72 hours, 96 hours, Day 7
  determine rate of organ failure (higher scores mean a worse outcome)
Plasma cytokines | baseline, 24 hours, 48 hours, Day 7
  IL-6, IL-4, IL-10, TNF-α, IL-1β/IL-1F2, CCL2/JE/MCP-1, IFN-gamma, IL-8/CXCL8
GDF-15, angiopoietin-2 | baseline, 24 hours, 48 hours, Day 7
  endothelial dysfunction
Hospital mortality | at hospital discharge, through study completion, an average 2 months
  death
Neurologic outcome | at hospital discharge, through study completion, an average 2 months
  Cerebral Performance Catergories scale

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Hoon Yang, MD, PhD, Principal Investigator — Department of Critical Care Medicine, Samsung Medical Center, Korea
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ko RE, Choi KH, Lee K, Jeon J, Jang HR, Chung CR, Cho YH, Park TK, Lee JM, Song YB, Hahn JY, Choi SH, Gwon HC, Yang JH. The effects of extracorporeal blood purification (oXiris(R)) in patients with cardiogenic shock who require VA-ECMO (CLEAN ECMO): a prospective, open-label, randomized controlled pilot study. Crit Care. 2025 Jun 20;29(1):255. doi: 10.1186/s13054-025-05495-4. PMID 40542431